CLINICAL TRIAL: NCT02101632
Title: Myorelaxant Effect of Bee Venom(BV) Topical Skin Application in Patients With Research Diagnostic Criteria/Temporomandibular Disorder Ia and Ib (RDC/TMD) Randomized, Double Blinded Study
Brief Title: Myorelaxant Effect of Bee Venom(BV) Topical Skin Application in Patients With RDC/TMD Ia and Ib
Acronym: BV/TMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Aleksandra Nitecka-Buchta, D.M.D., Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2012/07/B/ST6/01238
Record Dates: First submitted 2014-03-25; First posted 2014-04-02 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Other Disorders of Muscle in Diseases Classified Elsewhere
Keywords: TMD; bee venom; muscle tension; muscle pain
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bee Venom (Experimental): Bee Venom Ointment 0,0005%
  Interventions: Dietary Supplement: Bee Venom Ointment
- Vaseline (Placebo Comparator): Vaseline ointment
  Interventions: Other: Vaseline Ointment

INTERVENTIONS:
Dietary Supplement: Bee Venom Ointment — 2 weeks
  Arms: Bee Venom
Other: Vaseline Ointment — 2 weeks
  Arms: Vaseline

SUMMARY:
Topical application of BV ointment in patients with Research Diagnostic Criteria/Temporomandibular Disorder 1a and 1b (RDC/TMD) in experimental group, compared to placebo (vaseline) in control group.Application was repeated 3 times a day, during 14 days. Surface electromyography (EMG) was used to measure masseter rest tonus and maximal voluntary contraction tonus. Pain intensity was also analysed in VAS scale. Effectiveness of BV was compared with placebo in masseter myofascial pain in patients with TMD

DETAILED DESCRIPTION:
The aim of the study was evaluation of myorelaxant action of bee venom(BV) ointment, comparing to placebo.Parallel group, randomized double blinded trial was performed, including 79 patients with painful RDC/TMD 1a and 1b. Muscle tension was measured twice (TON1 and TON2) in rest muscle tonus (RMT) and maximal muscle contraction (MMC) on both sides right and left, with Easy Train Myo EMG (Version 3.1). Pain intensity was also analysed in VAS scale

ELIGIBILITY:
Inclusion Criteria:

* RDC/TMD 1a and 1b
* agreement to participate in the experimental study

Exclusion Criteria:

* bee venom allergy
* hyperactivity on bee products
* positive anamnesis of anaphylactic reaction after bee bites
* skin wounds with skin surface discontinuation
* RDC/TMD 2 and 3

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Masseter muscle tension | 2 weeks
  Masseter muscle tension at rest and in maximal voluntary contraction, electromyographic measurement [V]

SECONDARY OUTCOMES:
Pain intensity of masseter muscle | 2 weeks
  Pain intensity evaluation after 2 weeks of physiotherapy in visual analoque scale (VAS) scale

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Baron, Prof, Study Chair — Medical University of Silesia
Locations (1):
- Department of TMD and Orthodontics Silesian Medical University, Zabrze, Poland

REFERENCES:
- [Background] Hellner M, Winter D, von Georgi R, Munstedt K. Apitherapy: usage and experience in german beekeepers. Evid Based Complement Alternat Med. 2008 Dec;5(4):475-9. doi: 10.1093/ecam/nem052. Epub 2007 Jun 30. PMID 18955222
- [Background] Wieckiewicz W, Miernik M, Wieckiewicz M, Morawiec T. Does propolis help to maintain oral health? Evid Based Complement Alternat Med. 2013;2013:351062. doi: 10.1155/2013/351062. Epub 2013 Jan 9. PMID 23365605
- [Background] Kwon YB, Lee HJ, Han HJ, Mar WC, Kang SK, Yoon OB, Beitz AJ, Lee JH. The water-soluble fraction of bee venom produces antinociceptive and anti-inflammatory effects on rheumatoid arthritis in rats. Life Sci. 2002 May 31;71(2):191-204. doi: 10.1016/s0024-3205(02)01617-x. PMID 12031688
- [Background] Son DJ, Lee JW, Lee YH, Song HS, Lee CK, Hong JT. Therapeutic application of anti-arthritis, pain-releasing, and anti-cancer effects of bee venom and its constituent compounds. Pharmacol Ther. 2007 Aug;115(2):246-70. doi: 10.1016/j.pharmthera.2007.04.004. Epub 2007 May 6. PMID 17555825
- [Background] Seo BK, Lee JH, Sung WS, Song EM, Jo DJ. Bee venom acupuncture for the treatment of chronic low back pain: study protocol for a randomized, double-blinded, sham-controlled trial. Trials. 2013 Jan 14;14:16. doi: 10.1186/1745-6215-14-16. PMID 23317340
- [Derived] Nitecka-Buchta A, Buchta P, Tabenska-Bosakowska E, Walczynska-Dragon K, Baron S. Myorelaxant effect of bee venom topical skin application in patients with RDC/TMD Ia and RDC/TMD Ib: a randomized, double blinded study. Biomed Res Int. 2014;2014:296053. doi: 10.1155/2014/296053. Epub 2014 Jun 24. PMID 25050337